CLINICAL TRIAL: NCT02932917
Title: MapMySmoke: Feasibility of a New Quit Cigarette Smoking Mobile Phone Application Using Integrated Geo-positioning Technology, and Motivational Messaging Within Primary Care Setting
Brief Title: MapMySmoke: Smoking Cessation App With Geospatial Capture
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of St Andrews (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Robert Schick, MASTS Senior Research Fellow, University of St Andrews
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XAP062
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Smoking; Cigarette Smoking; Smoking, Tobacco
MeSH Terms: conditions — Smoking; Cigarette Smoking; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MapMySmoke (Experimental): All patients in the study will use the MapMySmoke app to document their smoking and craving behavior
  Interventions: Device: MapMySmoke

INTERVENTIONS:
Device: MapMySmoke — Each patient in the study arm will download and install the MapMySmoke app to record all of their smoking and craving events. The app will generate a quantitative summary of their smoking behavior during a pre-quit phase, and will provide dynamic text support messages during the post-quit phase. The app will also capture spatial details of any relapse events during the post-quit phase.

SUMMARY:
Place-based cues can be an important trigger of smoking behavior, therefore the investigators wish to learn more about the influence of the built environment on individual smoking behavior. This is to facilitate dynamic support during the post-quit phase. MapMySmoke is a mobile phone application that enables the capture of spatial data during smoking and craving events. These data will be used to create individualized support plans via the app.

DETAILED DESCRIPTION:
Investigators know that place-based cues play an important role in the triggering of smoking events, and even in relapse events. It follows that providing individual smokers with spatially explicit and temporally dynamic intervention messages may support smoking cessation attempts.

The investigators have built a mobile phone application-MayMySmoke-that allows individuals to capture each smoking event at the times and places they occur, and tag the events with qualitative metadata. The app also allows individuals to document and describe craving events. The goal of the app is first to understand an individual's smoking profile, and second to support them with dynamic text messages.

The investigators are deploying the app in a clinical setting-the United Kingdom's National Health Service, within the Fife region of Scotland. Using two feasibility studies of increasing size, the investigators are attempting first to get initial feedback on the app, and then to improve the app and deploy it across a broader community of smokers.

Though the app is targeted to smoking behavior, it is possible to extend it to include other negative health behaviors that may have a spatial component.

ELIGIBILITY:
Inclusion Criteria:

* National Health Service (Fife) Patients
* Self-reported tobacco smoker
* Stated intention to quit smoking
* English speaker

Exclusion Criteria:

* Mental illness
* learning difficulty

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Continued use of the MapMySmoke App as Assessed by Monitoring Individual Anonymized Data Feeds on the Server | 1 year
  The investigators will determine, via the data feed to the server, if patients continue to use the app during the pre- and post-quit phase

SECONDARY OUTCOMES:
Number of Patients Using the App Who Are Abstinent from Smoking As Assessed by Follow-up Survey | 4 weeks
  The investigators will determine via survey if patients have maintained their quit attempt
Number of Patients Using the App Who Are Abstinent from Smoking As Assessed by Follow-up Survey | 3 months
  The investigators will determine via survey if patients have maintained their quit attempt

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Schick, PhD, Principal Investigator — University of St Andrews

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schick RS, Kelsey TW, Marston J, Samson K, Humphris GW. MapMySmoke: feasibility of a new quit cigarette smoking mobile phone application using integrated geo-positioning technology, and motivational messaging within a primary care setting. Pilot Feasibility Stud. 2017 Jul 14;4:19. doi: 10.1186/s40814-017-0165-4. eCollection 2018. PMID 28725452